CLINICAL TRIAL: NCT07145099
Title: The IMPACT Study: A Randomized Controlled Trial of Individualized Management Post Ventral Hernia Repair (VHR) Utilizing Abdominal Core Therapy for Enhanced Recovery and Health Outcomes
Brief Title: The IMPACT Study: Personalized Physical Therapy for Better Recovery and a Stronger Core After Hernia Surgery
Acronym: IMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iRiSIDPending
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Ventral Hernia; Ventral Incisional Hernia; Post Operative Pain
Keywords: Physical Therapy; Rehabilitation; Economic Impact
MeSH Terms: conditions — Hernia, Ventral; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PT Group (Experimental): Initial Protocol (Post-Randomization): Participants will receive foundational instructions like usual care, including:
  Binder Use: Guidance on abdominal binder use.
  Lifting Precautions: Instruction on safe lifting techniques to protect the healing abdominal wall.
  Gradual Return to Activities: Advice on progressively re-engaging in daily activities.
  Tailored Physical Therapy Sessions (6 Sessions): Following the initial phase, participants will undergo 6 structured PT sessions. The progression and focus of these sessions will be individualized based on the participant's Oswestry Disability Index (ODI) score and Pelvic Floor Distress Inventory-20 (PFDI-20) score.
  Interventions: Other: PT Group
- Usual Care (Active Comparator): Protocol: Participants in this group will receive standard post-operative care instructions, which include:
  Binder Use: Guidance on the appropriate use of an abdominal binder.
  Lifting Precautions: Instruction on safe lifting techniques to protect the healing abdominal wall.
  Gradual Return to Activities: Advice on progressively re-engaging in daily activities.
  Follow-up: Participants will continue with usual care (no PT intervention) after the initial 12 weeks until the final assessment at Testing Session 2 (12 weeks post-operatively).
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: PT Group — Exercise, Manual Therapy, and education
  Arms: PT Group
Other: Usual Care — Education
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety, and cost-effectiveness of a tailored physical therapy (PT) intervention targeting Abdominal Core Health components in patients recovering from ventral hernia repair. The study focuses on patients aged 18-75 diagnosed with a ventral transverse hernia between 4 cm and 10 cm, scheduled for elective Ventral Hernia Repair (VHR).

The main questions it aims to answer are:

* Will tailored PT significantly improve abdominal core strength, biomechanical stability, and functional mobility compared to usual care at 3-months post-surgery?
* Will tailored PT lead to higher patient-reported quality of life and satisfaction scores, with a lower incidence of post-operative complications such as bowel obstruction and pelvic floor dysfunction over a 1-year follow-up?
* Will tailored PT result in decreased healthcare utilization, leading to overall cost savings or neutrality compared to usual care over the first year after VHR?

Researchers will compare the tailored physical therapy group to a usual care group to see if the tailored intervention leads to significant improvements in clinical efficacy, patient outcomes, and cost-effectiveness.

Participants will:

* Be randomly assigned to either the Usual Care Group or the PT Group.
* If in the Usual Care Group, receive standard post-operative instructions for 12 weeks, including guidance on binder use, safe lifting, and gradual return to activities.
* If in the PT Group, receive foundational post-operative instructions for the first 2 weeks (similar to usual care). Undergo 6 structured and individualized PT sessions over 10 weeks if in the PT Group, with progression based on Oswestry Disability Index (ODI) and Pelvic Floor Distress Inventory-20 (PFDI-20) scores, including Symptom Modulation, Movement Control, Functional Optimization, or Impairment-Based interventions.

Participants undergo data collection at 2 weeks, 12 weeks, and 1 year post-operation, including imaging, functional mobility tests, pain scales, patient-reported outcomes, physical measurements, and tracking of complications and healthcare utilization. Participate in semi-structured interviews after the 12-week assessment to provide qualitative insights into their experiences and perceived barriers/facilitators.

DETAILED DESCRIPTION:
The overarching goal of this project is to evaluate the efficacy, safety, and cost-effectiveness of a tailored physical therapy (PT) targeting Abdominal Core Health (ACH) components in patients recovering from ventral hernia repair (VHR). Specifically, we aim to:

Evaluate the clinical efficacy of tailored PT in improving abdominal core strength, biomechanical stability, and functional mobility. Hypothesis: Participants receiving the personalized PT intervention will demonstrate significant improvements in core strength, biomechanical parameters, and functional performance, compared to usual care at 3-months post-surgery. Objectives: 1.1. Measure changes in ultrasound-assessed abdominal muscle thickness (rectus abdominis, oblique and transversus abdominis muscles) and infra-sternal angle from baseline to 3-months post-surgery in both groups. 1.2. Quantify improvements in functional mobility via the 6-minute walk test and 30-second sit-to-stand test at 3-months post-surgery for all participants. 1.3. Compare incidence and severity of movement-related pain using validated pain scales between groups at 3-months.

Assess the impact of the tailored PT program on patient-reported outcomes and clinical complication rates. Hypothesis: Participants undergoing the tailored PT will report higher quality of life and satisfaction scores, with a lower incidence of post-operative complications such as bowel obstruction and pelvic floor dysfunction over a 1-year follow-up. Objectives: 2.1. Collect and compare patient-reported quality of life metrics and satisfaction with recovery scores at 3-months and 1-year post-surgery. 2.2. Track and compare the incidence of common post-VHR complications between groups over a 1-year follow-up period through medical record review and semi-structured interviews.

Elucidate mechanisms underlying post-VHR recovery and validate sensitive clinical measures for individualized treatment. Hypothesis: Changes in core biomechanics will positively associate with improvements in functional mobility and symptom reduction. Furthermore, quantitative measures will serve as reliable tools for monitoring recovery progress and guiding individualized treatment. Objectives: 3.1. Conduct correlation analyses between changes in biomechanical measures (Aim 1) and improvements in functional mobility and patient-reported outcomes (Aim 2) to identify key recovery pathways. 3.2. Evaluate the reliability and responsiveness of novel and existing quantitative measures (e.g., infra-sternal angle, abdominal circumference, pressure pain thresholds) as indicators of recovery progress and predictors of long-term outcomes.

Determine the cost-effectiveness of the personalized PT intervention compared to usual care. Hypothesis: The tailored PT will result in decreased healthcare utilization-fewer rehospitalizations, complications, and medication use over the first year after VHR-leading to overall cost savings or neutrality, supporting its integration into standard post-VHR care. Objectives: 4.1. Quantify and compare healthcare resource utilization (e.g., rehospitalizations, emergency department visits, specialist consultations, medication use) between groups over a 1-year follow-up. 4.2. Perform a comprehensive cost-effectiveness analysis from a healthcare system perspective, integrating direct and indirect costs with patient outcomes, to calculate the incremental cost-utility ratio of the intervention. 4.3. Conduct a qualitative assessment of patient and provider perceptions regarding the barriers and facilitators to intervention adherence and adoption, informing future implementation strategies.

Study Design and Approach: This research will be conducted as a Randomized Controlled Trial.

Selection and Justification of Intervention's Dose, Frequency, and Administration

The tailored PT intervention is designed as a structured, individualized program spanning 10 weeks of active therapy sessions, following an initial 2-week observation period post-randomization. This approach is rooted in contemporary understanding of abdominal core biomechanics and neuromuscular control, addressing the complex, multi-system nature of ACH. Current post-operative management for VHR often relies on general activity restrictions without comprehensively addressing these multi-system components, leading to potential complications and diminished functional capacity. The intervention's administration is highly personalized, adapting to the patient's evolving clinical status and specific needs as assessed by validated outcome measures:

Initial Protocol (Post-Randomization): For the first two weeks, participants in the PT group will receive foundational post-operative instructions similar to usual care, which include guidance on abdominal binder use and safe lifting techniques.

Tailored Physical Therapy Sessions (6 Sessions): Following this initial phase, participants will undergo six structured physical therapy sessions. The progression and specific focus of these sessions will be dynamically individualized based on the participant's ODI score and PFDI-20 score, which are reassessed prior to every session.

This individualized, adaptive dosing and administration protocol is justified by its alignment with the latest advancements in the Treatment-Based Classification system for low back pain, which has shown to result in improved outcomes through subgroup-matched treatments.This contrasts with traditional generalized recommendations, ensuring a patient-centered approach that directly addresses the unique biomechanical, physiological, and psychosocial profiles of individuals recovering from VHR.

Pelvic floor physical therapy plays a crucial role in the management of individuals with abdominal wall injuries such as diastasis recti, with studies demonstrating effectiveness of pelvic floor muscle training and core strengthening on inter-rectus distance and restoring function. Additionally, pelvic floor physical therapists are uniquely qualified to assess and treat coexisting pelvic floor dysfunction in those with abdominal wall injuries such as urinary incontinence and pelvic pain. This protocol provides comprehensive physical therapy treatment that addresses the integrated function of the musculature of the abdominal cavity, including the diaphragm, abdominals, lumbosacral, and pelvic floor muscles.

Sample Size: Sample size was calculated using the American Hernia Society Quality of Life (AHS-QC) outcome, a 0-100 point scale measuring patient quality of life after the operation. Based on prior studies, for the purposes of sample size estimation the mean AHS-QC score for the control group was assumed to be 47.6, with the treatment group possessing a mean AHS-QC score of 37.6, representing an approximately 20% reduction in score and a total effect size of 10.25 The standard deviation for both groups was assumed to be 15.6. Seeking to achieve 80% power in a two-sided two-sample t-test for difference in group means with a chosen significance level of 0.05, it was found that 40 patients were needed in each group, for 80 total, to achieve the desired power level. Assuming a combined loss to follow-up and incomplete response rate of 20%, it was determined that 100 patients should be the target enrollment of the study.

A sample of at least 10 participants each from the intervention and control group will be recruited for semi-structured interviews to meet sufficient informational power based on the standard five-dimensional approach for qualitative studies.

To answer the primary hypothesis, data will be collected on bowel obstruction occurrence rate, incidence of spine/pelvic floor diagnosis, pain intensity, patient-reported outcomes measures including the PFDI-20, AHS-QC, and ODI, functional outcomes measured by the 30-second sit-to-stand test and the 6-minute walk test (6MWT)

To assess the secondary hypothesis regarding biomechanical changes, dependent variables will include infra-sternal angle, abdominal circumference, abdominal muscle hypertrophy, pressure pain threshold, and two-point discrimination which will be measured by a trained and licensed physical therapist.

Qualitative Data: To address the secondary hypothesis on patient experience and satisfaction, semi-structured interviews will be conducted after the 12-week post-operative assessment. These sessions will include participants from both the PT and usual care groups in separate sessions. The interviews will explore patient perceptions of their post-operative care, their experiences with the PT intervention, and perceived benefits compared to standard care, providing rich qualitative data to complement quantitative satisfaction measures. Interview prompts and qualitative codes will be developed a priori, guided by the biopsychosocial model framework, and prior qualitative work on standard VHR and patient attrition in outpatient physical therapy. Interviews will be audio recorded and transcribed.

Economic Evaluation: The study will collect specific data on the costs associated with both groups over a 1-year period following the operation. This will include the direct costs of the physical therapy sessions (cost per session) for the intervention group, as well as healthcare utilization costs for both groups. These costs would then be compared against the value of the outcomes achieved (quantitative DVs).

Statistical Analysis Plan

Descriptive statistics such as means, medians, counts, and proportions will be calculated for each outcome and relevant cohort covariate.

To assess the primary hypothesis, a two-sample two-sided t-test will be employed to assess the mean difference in AHS-QC score between the treatment and control groups, with the test being performed at the 0.05 level. For other primary and secondary outcomes, point estimates along with 95% Wald confidence intervals for difference between the treatment and control groups will be calculated to present evidence of other between-group differences without a formal hypothesis test requiring adjustment for multiplicity.

In the analysis of each individual outcome, patients will be excluded from the analysis if they possess missing or incomplete measures of that outcome, with missingness assumed to be missing completely at random using Little's test and implementing an intent-to-treat analysis. Multiple imputation in R will be used if there happens to be a larger than expected amount of missing data (e.g., greater than 5%).

In the cost-utility analysis, clinical effectiveness will be measured at 1-year follow-up. A probabilistic sensitivity analysis will be conducted using the bootstrap method with 1000 replications. Results of the cost-utility analysis will be reported in accordance with best-practice standards.

Qualitative data will be analyzed via directed content analysis. Two independent raters will conduct qualitative coding (using independent thoughts as the unit of analysis), inter-rater reliability (Gwet's AC1 statistic) will be calculated, and all discrepancies will be resolved by consensus. Codes that include substantial thought units as agreed upon by both independent raters will be identified as themes. Themes will be summarized by group to understand differences in patient experience and impacts of the intervention as compared to the standard level of care. All qualitative methods will be conducted and reported in accordance with the consolidated criteria for reporting qualitative research.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18-75.
* Diagnosed clinically or via objective testing by a surgeon with a ventral transverse hernia >4 cm and <10 cm.
* Scheduled for elective surgical correction of a non-recurrent, primary or incisional ventral hernia.
* Independent functional status.

Exclusion Criteria:

* Individuals currently receiving or who have received PT within the last 30 days.
* Individuals currently using an assistive device for ambulation.
* Individuals diagnosed with a neurologic disorder will be excluded.
* History of or plan for Botox injection or muscle release related to the hernia.
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal Hernia Surgery Quality of Life Questionnaire | 2, 12, and 52 weeks.
  a validated patient-reported outcome measure assessing the impact of abdominal wall hernias and their repair on various aspects of quality of life. Scores are typically summed 0-100 with higher scores better.

SECONDARY OUTCOMES:
Bowel Obstruction Occurrence Rate | 52 weeks.
  The proportion or percentage of patients in each group who experience a bowel obstruction within the 1-year follow-up period.
Incidence of Spine/Pelvic Floor Diagnosis | 52 weeks.
  The number of new diagnoses of spine or pelvic floor conditions occurring in each group during the 1-year follow-up period.
Pain Intensity (SF-MPQ-2) | 2, 12, and 52 weeks.
  Pain intensity as measured by the Short-Form McGill Pain Questionnaire-2, a multidimensional pain assessment tool providing scores for continuous, intermittent, neuropathic, and affective pain. Scored between 0-220 with higher scores having more pain.
Pain Intensity (NPRS) | 2, 12, and 52 weeks.
  Pain intensity as rated by the Numerical Pain Rating Scale, typically a 0-10 scale where 0 represents "no pain" and 10 represents "worst imaginable pain."
PROMIS Pain Interference | 2, 12, and 52 weeks.
  Assesses the impact of pain on physical, mental, and social functioning, as well as sleep and enjoyment of life. a 5-point scale with 6 items with a highest possible raw score of 0- 30. Higher scores are worse.
30-Second Sit-to-Stand Test | 2, 12, and 52 weeks.
  The number of times a patient can rise to a full standing position from a seated position in 30 seconds, assessing lower extremity strength and functional mobility.
6-Minute Walk Test (6MWT) | 2, 12, and 52 weeks.
  The total distance (in meters or feet) a patient can walk at a comfortable pace over 6 minutes assessing exercise tolerance and functional capacity.
Infra-sternal Angle | 2, 12, and 52 weeks.
  The angle formed by the left and right costal margins at the xiphoid process, reflecting rib cage orientation and potentially core stability. Measured in degrees.
Abdominal Circumference | 2, 12, and 52 weeks.
  The measurement of the circumference around the abdomen, typically taken at a specific anatomical landmark (e.g., umbilicus), reflecting abdominal size and potentially muscle changes. Measured in cm or inches.
Abdominal Muscle Hypertrophy | 2, 12, and 52 weeks.
  Change in the size or thickness of specific abdominal muscles (e.g., rectus abdominis, obliques) as measured by imaging techniques (ultrasound). Measured in units of length or area.
Pressure Pain Threshold | 2, 12, and 52 weeks.
  The minimum amount of pressure applied to a specific point that elicits a sensation of pain, indicating tissue sensitivity. Measured in units of pressure (kg).
Two-Point Discrimination | 2, 12, and 52 weeks.
  The minimum distance between two simultaneously applied points that can be perceived as distinct stimuli, assessing tactile spatial acuity. Measured in millimeters.

OTHER OUTCOMES:
Complications & Healthcare Utilization | 52 weeks
  Tracked via medical record review and structured interviews.
Economic Analysis | 52 weeks
  Direct costs of PT sessions and healthcare utilization costs (e.g., physician visits, hospital admissions, medications, complication management) will be systematically collected from medical records and billing data. Indirect costs such as lost productivity or time away from work, will be estimated using patient-reported employment status and time off work, valued using average regional wage data.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Keating, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with reasonable request to PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon the end of the study.
Access Criteria: Email